CLINICAL TRIAL: NCT01786200
Title: Pilot Study to Investigate the Physiological Effects Associated With Down-regulation of Host-tumour Inflammatory Responses in Colon Cancer
Brief Title: Physiological Effects of Altering Cancer-related Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Academy of Medical Sciences (Ambiguous); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GN12SU401; 12736 (Registry Identifier: UKCRN)
Record Dates: First submitted 2013-01-29; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Colon Cancer
Keywords: colon; cancer; NSAID; inflammation
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms; Inflammation | interventions — Aspirin; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspirin (Active Comparator): 20 patients randomised to aspirin 75mg PO once daily
  Interventions: Drug: Aspirin
- Ibuprofen (Active Comparator): 20 patients randomised to ibuprofen 400mg PO three times daily
  Interventions: Drug: Ibuprofen
- Control (No Intervention): 20 patients randomised to receive no treatment

INTERVENTIONS:
Drug: Aspirin
  Arms: Aspirin
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
This prospective pilot study will examine whether the previously reported effects of NSAIDs on colorectal cancer may be modulated through alterations in tissue gene expression, up regulation of local immune cell infiltrates or down-regulation of the systemic inflammatory response.

DETAILED DESCRIPTION:
Bowel cancer is the second commonest cause of death from cancer in the UK. Of patients who have an apparently curative operation, half unfortunately suffer disease recurrence and die before 5 years. Clearly more research is required to improve outcomes in this condition. Most current research focuses on antitumour strategies, however the reaction of the patient (host) to the tumour is also important. The host inflammatory responses to the cancer are likely to represent part of this host-tumour relationship. Inflammation plays an important role in predicting patients who will die. Currently it is not known whether antiinflammatory drugs have any effect on cancer related inflammation detected in the blood or in/around the tumour.

Aims: We hope to demonstrate that tumour related inflammation in bowel cancer can be altered using anti- inflammatory drugs. This may form the rationale for the use of antiinflammatory drugs to improve prognosis in colorectal cancer patients undergoing surgery.

Methods: This pilot study will investigate whether simple antiinflammatory drugs can alter markers of inflammation both in the blood and in/around the tumour. Patients having bowel cancer surgery will be prescribed one of two anti-inflammatory drugs (aspirin 75mg once daily or ibuprofen 400mg three times daily) for 2 to 3 weeks prior to their operation. Blood and tumour samples before and after the treatment will be analysed.

If the study's aims are met and cancer-related inflammation can be altered prior to surgery, then a larger scale drug trial will be proposed to demonstrate reduced cancer recurrence and improved survival.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 75 years old
* histologically confirmed colon cancer
* evidence of systemic inflammation (C-reactive protein >10mg/l)
* candidate for elective primary curative resection

Exclusion Criteria:

* Age <18yrs or >75yrs
* emergency presentation
* rectal cancer
* distal metastatic disease at presentation
* provision of neo-adjuvant chemo-radiotherapy
* long-term use of aspirin or anti-inflammatory medications (NSAIDS, or steroids
* hypersensitivity to product or excipients or evidence of previous hypersensitivity reactions such as asthma, rhinitis, angioedema or urticaria in response to aspirin, ibuprofen or other NSAID
* intolerance of NSAIDs/ aspirin due to allergy or side effects
* active peptic ulcer disease
* previous history of recurrent gastrointestinal bleeding or bleeding/perforation secondary to previous NSAID use
* previous treatment for gastrointestinal cancer
* alcohol excess (above recommended guidelines)
* chronic renal impairment
* moderate to severe heart failure
* hepatic impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Klintrup-Makinen immune score | Approx 4 weeks (post-treatment and surgery)
  To evaluate the local inflammatory effects associated with down-regulation of the systemic inflammatory response prior to curative surgery as measured by Klintrup-Makinen immune score

SECONDARY OUTCOMES:
Systemic inflammatory response | Approx 4 weeks (post-treatment and surgery)
  Comprehensive assessment of the systemic inflammatory response prior to curative surgery as measured by C-reactive protein (CRP), differential white cell count, albumin and cytokines (IL-1, 6,8 and 10, TNF-alpha)
Assessment of gene inflammatory profile | Approx 4 weeks (post-treatment and surgery)
Local inflammatory response | Approx 4 weeks (post-treatment and surgery)
  Immunohistochemical analysis of immune cells infiltrates in colonic and tumour tissue will be performed quantitatively. Cell surface antigens evaluated include CD4+, CD8+, CD68+, CD45RO+ and FOXP3+.

CONTACTS AND LOCATIONS:
Overall Officials: Campbell Roxburgh, Principal Investigator — University of Glasgow
Locations (1):
- Glasgow Royal Infirmary - Walton Building, Glasgow, United Kingdom